CLINICAL TRIAL: NCT03370250
Title: Immediate Breast Reconstruction With Free Greater Omentum for Luminal Breast Cancer Patients
Brief Title: Immediate Breast Reconstruction With Free Greater Omentum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20162047-1
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Breast Reconstruction
Keywords: immediate breast reconstruction; free greater omentum; breast-conserving surgery; luminal breast cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Luminal subtype breast cancer, accounting for 70 to 80% of all breast cancers, has been reported to be associated with good prognosis. However, for the patients with large mass or worse mass position, free greater omentum transplantation may provide a new option for breast reconstruction.

DETAILED DESCRIPTION:
Breast-conserving surgery, laparoscopic greater omentum harvest and vascular anastomosis was carried out orderly. The omentum was harvested laparoscopically, following breast-conserving surgery . Following the remove of resected omentum, the harvested greater omentum was poured by ice protection fluid from right gastric omentum artery. Besides, right arteriovenous vein of stomach omentum was dissected carefully under microscope. When operation started, front latissimus dorsi was separated from subaxillary incision, as well as the right thoracic dorsal artery and accompanying vein. Separated greater omentum was put on the subcutaneous deficient site of right breast incision and vascular pedicle was pulled through tunnel, reaching to the axillary incision. Under the help of microscope, vascular anastomosis between right stomach omentum arteriovenous and right thoracic dorsal arteriovenous was proceeded. Consequently, greater omentum was filled to shape the reconstructed breast. Finally, drainage tube and drainage strip were left at subcutaneous and subaxillary incision, respectively.

ELIGIBILITY:
Inclusion Criteria:

- Patient aged 18 -60 years Patient diagnosed with luminal breast cancer No neoadjuvant chemotherapy previously No distant metastasis Suitable for breast conserving surgery Willing and able to give written informed consent to participate in the study including all follow-up examinations

Exclusion Criteria:

- Participate in another clinicaltrial Bilateral lesions Pregnancy or lactation Greater omentum unable to extract or insufficient omentum Other surgical contraindication

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The research team selected the patients diagnosed with breast cancer and classified as luminal subtype who received one-sided therapeutic mastectomy and breast reconstruction with free omentum flap between January 23, 2015 and December 6, 2017
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
severe related complication | 1 year after surgery
  Serious adverse effect occur within 1 years after implantation

SECONDARY OUTCOMES:
cosmetic outcome | 6 months after surgery
  Four-point scale was formulated to evaluate the cosmetic score as excellent (size and shape of recon-structed breast are identical to the original breast); good (deformity of the reconstructed breast in-volved less than 1/4 of the original breast; fair (deformity of the reconstructed breast involves less than 1/4-1/2 of the original breast); and poor (breast deformity involves more than 1/2 of the original breast)
greater omentum survival | 2 and 5 years after surgery
  At each follow up time point the proportion of patients with omentum transplantation will be estimated.
Patient satisfaction | 6months, 1 and 2 years after surgery
  Patients also rate their level of satisfaction, with the help of a numeric rating scale (NRS: 0-10), in terms of how the outcome met up to their preoperative expectations of the arthroplasty. Finally, they will be asked whether - with their current knowledge of the outcome - they would again choose the operation if they found themselves in similar circumstances to those which prevailed preoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China